CLINICAL TRIAL: NCT03002246
Title: Automated Fetal Weight Estimation: A Multicenter Validation Using Fractional Limb Volume
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Samsung Medison Co., Ltd. (Unknown); Beijing Obstetrics and Gynecology Hospital (Other); Frauenklinik der Diakonischen Dienste Hannover (Unknown); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Wesley Lee, Dr. Wesley Lee, Baylor College of Medicine
Other Study IDs: H-39343
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Birth Weight; Fetal Growth Retardation; Fetal Weight; Fetal Macrosomia
MeSH Terms: conditions — Birth Weight; Fetal Growth Retardation; Fetal Weight; Fetal Macrosomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Average for Gestational Age: This cohort will include a sample size of 90 subjects. Fetuses will have an estimated fetal weight greater than 10th percentile and less than 90th percentile based on clinical ultrasound assessment. This cohort will receive an ultrasound examination 4-7 days before their delivery.
  Interventions: Other: Ultrasound Examination
- Large for Gestational Age: This cohort will include a sample size of 30 subjects. Fetuses will have an estimated fetal weight greater than 90th percentile based on clinical ultrasound assessment.This cohort will receive an ultrasound examination 4-7 days before their delivery.
  Interventions: Other: Ultrasound Examination
- Small for Gestational Age: This cohort will include a sample size of 30 subjects. Fetuses will have an estimated fetal weight less than 10th percentile based on clinical ultrasound assessment.This cohort will receive an ultrasound examination 4-7 days before their delivery.
  Interventions: Other: Ultrasound Examination

INTERVENTIONS:
Other: Ultrasound Examination — Research volunteers will be invited to have a 2D/3D ultrasound research scan 4-7 days from delivery.This ultrasound scan will take approximately 30 minutes to complete.

SUMMARY:
This trial is a collaborative study between 4 sites worldwide. A total of 600 research subjects will be enrolled. We will investigate the validity of using 5D Limb Volume software to improve on estimated fetal weight predictions over a broad range of gestational ages. The purpose is to compare the accuracy and precision of birth weight predictions based on this new technology as compared to the current 2D birth weight prediction models.

DETAILED DESCRIPTION:
Ultrasound has been used for over 20 years to estimate fetal weight prior to birth. Sometimes this estimation is not always similar to what the baby actually weighs. In addition to the regular measurements taken at routine ultrasound exams, 3D ultrasound of the baby's arm and leg soft tissue may give us more precise information on how much the baby weighs. This measurement is called fractional limb volume. Fractional limb volume (FLV) is a soft tissue measurement of the arm or thigh that can be used to evaluate body composition. This measurement mostly reflects the fat and muscle development with a small amount of bone.

The recent introduction of 5D Limb Volume software (Samsung, Seoul, Korea) now makes it possible to efficiently and reproducibly measure semi-automated FLV using a computer guided technique.

Subjects will receive one ultrasound scan 4-7 days before their delivery. Both 2D and 3D measurements will be taken. These measurements will then be used to estimate fetal weight. We will compare estimated weight to actual birth weight in order to determine the accuracy and precision of the 5D Limb Volume technology. This data may also be used to develop new weight estimation models that could provide better accuracy and/or precision than what is currently provided using published methods.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women (28-42 weeks) within 4-7 days of delivery
2. Planned delivery at the collaborating hospital where the fetal US scan was performed
3. Body mass index at first official prenatal appointment below 35.0 kg/M2
4. Firm US dating criteria (early crown-rump length < 14 weeks gestational age)

Exclusion Criteria:

1. Presence of technical factors (e.g. obesity) that make it difficult to visualize fetal structures
2. Oligohydramnios determined by amniotic fluid index less than 5cm
3. Fetal distress or unstable maternal condition
4. Structural or chromosomal fetal anomalies

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between 28-42 weeks gestation. Fetuses will be either small for gestational age (estimated fetal weight < 10%), average for gestational age, or large for gestational age (estimated fetal weight > 90%).
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Comparison Between 5D Limb Vol and 2D Birth weight Prediction | Feb 2017 -Feb 2018
  Compare the accuracy and precision of BW predictions based on 5D Limb Vol technology in pregnant women as compared to 2D BW prediction models

SECONDARY OUTCOMES:
Birth weight Predictions in Suspected Growth Abnormalities | Feb 2017 - Feb 2018
  Characterize the performance of BW predictions based on 5D Limb Vol technology in pregnant women with suspected growth abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Lee, MD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kang L, Wu QQ, Sun LJ, Gao FY, Wang JJ. Predicting fetal weight by three-dimensional limb volume ultrasound (AVol/TVol) and abdominal circumference. Chin Med J (Engl). 2021 Apr 20;134(9):1070-1078. doi: 10.1097/CM9.0000000000001413. PMID 33883411